CLINICAL TRIAL: NCT05998018
Title: Randomized Study of the pdSTIM™ System (Phrenic Nerve to Diaphragm STIMulation) in Failure to Wean Mechanically Ventilated Patients
Brief Title: Randomized Study of the pdSTIM™ System in Failure to Wean Mechanically Ventilated Patients
Acronym: ReInvigorate
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment was temporarily paused to allow for protocol evaluation and planned modifications.
Sponsor: Stimdia Medical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIP0002
Record Dates: First submitted 2023-08-11; First posted 2023-08-18 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-05

CONDITIONS: Neuromodulation; Phrenic Nerve Stimulation; Ventilator Induced Diaphragm Dysfunction; Mechanical Ventilation Weaning
Keywords: Mechanical Ventilation; Phrenic Nerve Stimulation; Neuromodulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- pdSTIM System Therapy (Experimental)
  Interventions: Device: pdSTIM System Therapy; Other: Conventional Medical Management
- Standard of Care (Active Comparator)
  Interventions: Other: Conventional Medical Management

INTERVENTIONS:
Device: pdSTIM System Therapy — Stimulate the phrenic nerves in synchrony with inspiratory cycles of the ventilator which exercises the diaphragm
  Arms: pdSTIM System Therapy
Other: Conventional Medical Management — Conventional medical management

SUMMARY:
This prospective, multi-center, randomized, controlled clinical trial is being conducted to evaluate the safety and efficacy of the pdSTIM System to facilitate weaning from mechanical ventilation through phrenic nerve stimulation. Potential subjects who are on mechanical ventilation for at least four days and have failed at least one weaning attempt will be considered for the study. Those enrolled will be randomized in a 1:1 manner between the treatment group that is standard of care with the pdSTIM System and a Control group, which is standard of care alone.

DETAILED DESCRIPTION:
The pdSTIM Pivotal Study (ReInvigorate Study) is a prospective, multicenter, randomized, controlled clinical study to evaluate the safety and efficacy of the pdSTIM System to facilitate weaning from mechanical ventilation through phrenic nerve stimulation. Potential subjects who are on mechanical ventilation for ≥ 96 hours (4 days) and have failed at least one weaning attempt will be considered for the study.

Those enrolled will be randomized in a 1:1 manner between a Treatment group that is standard of care with the pdSTIM System and a Control group that is standard of care only. For the Treatment group, stimulation therapy with pdSTIM will occur daily until the subject is successfully removed from mechanical ventilation or the 30-Day follow-up visit, whichever is sooner. All randomized subjects will be followed to 60 (± 7) days post randomization. Total subject participation will be no longer than 67 days.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is 18 years or older.
2. Subject, or subject's Legally Authorized Representative, understands study requirements, study visits, and is willing and able to provide written informed consent prior to study specific procedures or testing.
3. Subject has been on mechanical ventilation for ≥ 96 hours prior to randomization (intubation or tracheostomy).
4. Subject has failed at least 1 weaning attempt (e.g., site directed spontaneous breathing trial(s) did not result in liberation).
5. At the time of enrollment, the subject is likely to be ventilated for an additional 48 hours, at minimum, in the opinion of the investigator.

Exclusion Criteria:

1. Subject has been on invasive mechanical ventilation for > 45 days.
2. Subject failed to wean due to pre-existing neurological or neuromuscular issues affecting the respiratory muscles (e.g., ALS, phrenic nerve paralysis, inflammatory muscle disease, underlying myopathy, myasthenia gravis, cervical spinal injury).
3. Subject's medical history, known anatomy or investigator's inability to visualize necessary anatomical landmarks that could prevent the safe placement of the pdSTIM leads.
4. Subject is at risk of significant hemorrhage or is currently receiving a full dose of systemic anticoagulation (e.g., IV heparin, high dose of subcutaneous heparin. Subjects on prophylactic anticoagulation or daily aspirin regimen on their own are not excluded unless other exclusion criteria apply).
5. Subject has an implant or external electrical device that may interact or interfere with the pdSTIM System (examples may include cardiac pacemaker, implantable defibrillator, vagal nerve stimulator, spinal cord stimulator, gastric stimulator, diaphragmatic stimulator).
6. Subject has been diagnosed and has been treated for neck cancer within the past 5 years or subject had any prior radiation treatment to the neck.
7. Subject currently has hemodynamic instability due to any cause (e.g., severe sepsis, hemorrhagic shock, or septic shock) with vasopressor support > 0.1 mg/kg/min of norepinephrine or epinephrine, or equivalent, or is actively being titrated.
8. Subject has a local infection at or around the proposed pdSTIM Lead insertion site.
9. Subject is neutropenic or has signs of significant immunocompromise. (Subjects intubated for respiratory failure due to COVID-19 are not excluded unless other exclusion criteria apply).
10. Subject has severe COPD as indicated by evidence of significant expiratory obstruction on the ventilator flow waveform or, where ventilator flow waveforms are not utilized, has a FEV1 ≤ 30%.
11. Subject has pre-existing severe chronic pulmonary fibrosis.
12. Subject has pleural effusion occupying greater than 1/3 of the pleural space on either side.
13. Subject is currently on or expected to begin neuromuscular blockades.
14. Subject is anticipating withdrawal of life support and/or shift to palliation as the goal of care with less than 6-months life expectancy.
15. Subject is known or suspected to be pregnant or lactating.
16. Subject is currently enrolled in or exited early from a) any investigational drug study or b) an investigational device study that may impact the ability to wean or is directly related to the lungs or diaphragm.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2023-09-29 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Time to Wean | Following completion of the 30-day follow-up by all available randomized subjects
  Assess time to successful weaning from mechanical ventilation for the subjects randomized to Treatment as compared to subjects randomized to Control
Assessment of Serious Adverse Events (SAEs) | Following completion of the 30-day follow-up by all available randomized subjects
  Assessment of Serious Adverse Events (SAEs) for the subjects randomized to Treatment as compared to subjects randomized to Control

SECONDARY OUTCOMES:
Mortality Rates | Following completion of the 30-day follow-up by all available randomized subjects
  Compare 30-day mortality rates of Treatment and Control subjects
Adverse Event Rates | Following completion of the 30-day follow-up by all available randomized subjects
  Compare adverse event rates for Treatment and Control subjects
Days on Mechanical Ventilation | Following completion of the 30-day follow-up by all available randomized subjects
  Compare number of days on mechanical ventilation from the date of randomization to removal of mechanical ventilation associated with successful weaning or Day 30, whichever comes first, for Treatment and Control subjects

OTHER OUTCOMES:
pdSTIM System Summary | Following completion of the 30-day follow-up by all available randomized subjects
  Summarize pdSTIM System characteristics, such as lead placement success rate, duration of procedure, waveforms of flow/pressure, and programmed parameters over time
Mean Change in Rapid Shallow Breathing Index (RSBI) | Following completion of the 30-day follow-up by all available randomized subjects
  Compare the mean change in Rapid Shallow Breathing Index from randomization to Day 30 or removal of mechanical ventilation, whichever comes first, for Treatment and Control subjects
Number of ICU Days | Following completion of the 30-day follow-up by all available randomized subjects
  Compare the number of ICU days from randomization to Day 30 or removal of mechanical ventilation, whichever comes first, for Treatment and Control subjects
Rate of Re-intubation | Following completion of the 30-day follow-up by all available randomized subjects
  Compare the rate of re-intubation following successful weaning for Treatment and Control subjects

CONTACTS AND LOCATIONS:
Overall Officials: Steven Conrad, MD,PhD, Principal Investigator — LSU Health Sciences Shreveport
Locations (21):
- United States (21):
  - University of South Alabama, Mobile, Alabama
  - Chandler Regional Medical Center, Chandler, Arizona
  - Abrazo West Campus, Goodyear, Arizona
  - HonorHealth Research Institute, Scottsdale, Arizona
  - Denver Health, Denver, Colorado
  - Grady Memorial Hospital, Atlanta, Georgia
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - University of Illinois Chicago, Chicago, Illinois
  - RML Specialty Hospital, Hinsdale, Illinois
  - University of Louisville, Louisville, Kentucky
  - Tulane University Medical Center, New Orleans, Louisiana
  - LSU Health Sciences Center at Shreveport, Shreveport, Louisiana
  - University of Michigan Health - West, Wyoming, Michigan
  - Northwell South Shore University Hospital, Bay Shore, New York
  - University at Buffalo, Buffalo, New York
  - Atrium Health Carolinas Medical Center, Charlotte, North Carolina
  - WakeMed Health, Raleigh, North Carolina
  - Forsyth Medical Center, Winston-Salem, North Carolina
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - St. David's Healthcare, Georgetown, Texas
  - Houston Methodist, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schaaf K, Mullin CM, Cunningham KW, Eaton J, Conrad SA. The ReInvigorate Study-phrenic nerve-to-diaphragm stimulation for weaning from mechanical ventilation: a protocol for a randomized pivotal clinical trial. Trials. 2024 Aug 2;25(1):519. doi: 10.1186/s13063-024-08355-8. PMID 39095923
- See also: Company Website — https://stimdia.com/